CLINICAL TRIAL: NCT06812754
Title: A Phase 2, Randomized, Placebo-controlled, 12-week, Double-blind Study to Assess the Efficacy and Safety of Fezolinetant 45 mg in Chinese Women Suffering From Moderate to Severe Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Confirm if Fezolinetant Helps Reduce Hot Flashes in Chinese Women Going Through Menopause
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2693-CL-0313; CTR20250084 (Registry Identifier: ChinaDrugTrials.org.cn)
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Hot Flashes
Keywords: ESN364; vasomotor symptoms; fezolinetant; VEOZAH™; menopause
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fezolinetant (Experimental): Participants will receive fezolinetant once daily for 12 weeks.
  Interventions: Drug: Fezolinetant
- Placebo (Placebo Comparator): Participants will receive matching placebo once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fezolinetant — oral
  Other Names: ESN364; VEOZAH™
  Arms: Fezolinetant
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
Hot flashes are the most common reason women going through menopause seek medical attention. Hormone replacement therapy, or HRT, is most often prescribed to treat hot flashes. However, HRT can't be used by all women or for as long as may be needed.

The goal of this study is to confirm if fezolinetant helps reduce hot flashes in Chinese women going through menopause. This study will also confirm the safety of fezolinetant and how well the women cope with (tolerate) the treatment. The women will take 1 tablet of the study medicine either fezolinetant or placebo once a day for up to 12 weeks. This is decided by chance alone. The placebo looks like fezolinetant but will not have any medicine in it.

Women that want to take part in the study will be given an electronic handheld device with an app to track their hot flashes and night sweats. The women will record this information before, during and after taking the study treatment. During the study, the women will visit the study clinic several times. At each visit they will be asked if they had any medical problems. The women will have general safety checks. At some visits, a breast ultrasound (mammogram), cervical smear, and ultrasound of the womb (uterus) may be done.

The last clinic visit will be 3 weeks after the women take their final tablet of the study medicine (fezolinetant or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index >/= 16 kg/m2 and </= 38 kg/m2 at screening visit.
* Participant must be seeking treatment or relief for vasomotor symptom(s) (VMS) associated with menopause and confirmed as menopausal per 1 of the following criteria at the screening visit:

  * Spontaneous amenorrhea for >/= 12 consecutive months
  * Spontaneous amenorrhea for >/= 6 months with biochemical criteria of menopause (follicle-stimulating hormone (FSH) > 40 IU/L); or
  * Having had bilateral oophorectomy >/= 6 weeks prior to the screening visit (with or without hysterectomy).
  * FSH > 40 IU/L if participants received hysterectomy but still have an ovary/ovaries.
* Within the 10 days prior to randomization, participant must have a minimum average of 7 moderate to severe hot flash(es) (HFs) (VMS) per day (data must be available for at least 7 of the last 10 days prior to randomization).
* Participant is in good general health as determined on the basis of medical history and general physical examination, performed at the screening visit; hematology and biochemistry parameters, pulse rate and/or blood pressure, and electrocardiogram (ECG) within the reference range for the population studied, or showing no clinically relevant deviations.
* Participant has documentation of a normal/negative or no clinically significant findings mammogram (or breast ultrasound) (e.g., < Breast Imaging-Reporting and Data System (BI-RADS) class 4; obtained at screening or within the prior 12 months of study enrollment). Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant mammographic findings.
* Participant is willing to undergo a transvaginal ultrasound (TVU) to evaluate the uterus and ovaries at screening and week 12 (end of treatment (EOT)), and for participants who are withdrawn from the study prior to completion, a TVU at the early discontinuation (ED) visit. This is not required for participants who have had a partial (supracervical) or total hysterectomy.
* Participant has documentation of a normal or not clinically significant Pap test (or equivalent cervical cytology) within the previous 12 months of study enrollment or at screening. This is not required for participants who have had a total hysterectomy.
* Participant has a negative urine pregnancy test at screening; this is not required for participants who have had a total hysterectomy.
* Participant has a negative serology panel [i.e., negative hepatitis B surface antigen (HBsAg) and negative hepatitis C virus antibody (HCVAb) screens] at screening.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has known substance abuse or alcohol addiction within 6 months of screening.
* Participant has a current malignancy, with exception of non-metastatic basal cell carcinoma of the skin.
* Participant has a history of malignancy with exceptions of at least 5 years post-treatment and without known recurrence.
* For participants with a uterus: Participant has an unacceptable result from the TVU assessment at screening, i.e., full length of endometrial cavity cannot be visualized or presence of a clinically significant finding.
* Participant has a history within the last 6 months of undiagnosed uterine bleeding.
* Participant has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine, or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Participant has a history of suicide attempt or suicidal behavior within the last 12 months or has suicidal ideation within the last 12 months (a response of "yes" to question 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale [C-SSRS]), or who is at significant risk to commit suicide at screening [visit 1].
* Participant has previously been enrolled in a clinical trial with fezolinetant or other neurokinin (NK) receptor antagonists.
* Participant uses a prohibited therapy (strong and moderate cytochrome P450 1A2 [CYP1A2] inhibitors, hormone replacement therapy (HRT), hormonal contraceptive or any treatment for VMS [prescription, over-the-counter, or herbal]) or is not willing to wash-out and discontinue use of such drugs for the full duration of study conduct.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has uncontrolled hypertension, defined as systolic blood pressure >/=140 mmHg or diastolic blood pressure as >/= 90 mmHg based on an average of 2 to 3 readings within the screening period.

  * Participants with a medical history of hypertension who are well controlled may be enrolled
  * Participants who do not meet these criteria may be re-assessed after initiation or review of antihypertensive measures
* Participant has active liver disease, jaundice, elevated liver aminotransferases (alanine aminotransferase (ALT) or aspartate aminotransferase (AST)), elevated total or direct bilirubin, elevated international normalized ratio (INR) or elevated alkaline phosphatase (ALP). Patients with mildly elevated ALT or AST up to 1.5 × upper limit of normal (ULN) can be enrolled if total and direct bilirubin are normal. Patients with mildly elevated ALP (up to 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Patients with Gilbert's syndrome with elevated total bilirubin (TBL) may be enrolled as long as hemolysis is ruled-out (i.e., direct bilirubin, hemoglobin and reticulocytes are normal).
* Participant has creatinine > 1.5 × ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula </=30 mL/min/1.73 m2 at screening.
* Participant has a positive result for human immunodeficiency virus (HIV) at screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant is unable or unwilling to complete the study procedures.
* Participant has a known or suspected hypersensitivity to fezolinetant or any components of the formulation used.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in the frequency of moderate to severe Vasomotor Symptoms (VMS) from baseline to week 12 | Baseline to Week 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day.

SECONDARY OUTCOMES:
Mean change in the frequency of moderate to severe VMS from baseline to each week up to week 12 | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day.
Mean change in the severity of moderate to severe VMS from baseline to week 12 | Baseline to Week 12
  The severity of VMS will be calculated using a weighted average of VMS events.
Mean change in the severity of moderate to severe VMS from baseline to each week up to week 12 | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  The severity of VMS will be calculated using a weighted average of VMS events.
Mean percent reduction in the frequency of moderate to severe VMS from baseline to each week up to week 12 | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate or severe VMS events per day. Mean percent reduction will be reported.
Percent reduction >/= 50% in the frequency of moderate to severe VMS from baseline to each week up to week 12 | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day. Percent reduction of >/= 50% will be reported.
Percent reduction at 100% in the frequency of moderate to severe VMS from baseline to each week up to week 12 | Baseline to Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day. Percent reduction of 100% will be reported.
Number of participants with Adverse Events (AEs) | Up to Week 15
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Change from baseline in endometrial thickness in post-menopausal participants | Baseline up to Week 12
  Endometrial thickness is a measure of how thick the lining of the uterus is. Endometrial thickness will be measured by transvaginal ultrasound (TVU).
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to Week 15
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to Week 15
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to Week 12
  Number of participants with potentially clinically significant ECG values.
Pharmacokinetics (PK) of Fezolinetant in plasma: Concentration | Up to Week 12
  Concentration will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of metabolite ES259564 in plasma: Concentration | Up to Week 12
  Concentration will be recorded from the PK plasma samples collected.
Change in serum concentrations of sex hormones | Baseline up to Week 15
  Sex hormone biomarker levels will be recorded from serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Astellas Pharma Global Development, Inc.
Locations (27):
- China (27):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Capital Medical University (CMU) - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Capital Medical University - Beijing Obstetrics and Gynecology Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangzhou Medical University - The Third Affiliated Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Maternal & Child Health Hospital, Shenzhen, Guangdong
  - Guangxi Medical University (GXMU) - Liuzhou Renmin Hospital, Liuchow, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Hainan Women and Children's Medical Center, Haikou, Hainan
  - The second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Zhuzhou, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Southeast University, ZhongDa Hospital, Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Jilin Province FAW General Hospital, Changchun, Jilin
  - Jinan Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - Shanxi Woman and Children Hospital, Taiyuan, Shanxi
  - The First hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/